CLINICAL TRIAL: NCT03874260
Title: A Multi-center, Randomized, Double-blind, Parallel Phase Ⅳ Study to Explore the Efficacy of Statin/Choline Fenofibrate Combination Therapy vs Statin Monotherapy in Patients With Inadequately Controlled TG Despite Receiving Statin Monotherapy
Brief Title: Cinical Trial to Explore the Efficacy of Statin/Choline Fenofibrate Combination Therapy vs Statin Monotherapy in Patients With Inadequately Controlled TG Despite Receiving Statin Monotherapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DWTF-401
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias | interventions — Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- statin / fenofibrate (Experimental): stable statin(rosuvastatin 10mg or atorvastatin 10mg or atorvastatin 20mg)+ choline fenofibrate 178.8mg / once a day, P.O
  Interventions: Drug: Fenofibrate
- statin / fenofibrate placebo (Placebo Comparator): stable statin(rosuvastatin 10mg or atorvastatin 10mg or atorvastatin 20mg) + choline fenofibrate placebo / once a day, P.O
  Interventions: Drug: Fenofibrate

INTERVENTIONS:
Drug: Fenofibrate — statin(rosuvastatin 10mg or atorvastatin 10mg or atorvastatin 20mg) + choline fenofibrate vs statin(rosuvastatin 10mg or atorvastatin 10mg or atorvastatin 20mg) + choline fenofibrate placebo / once a day, P.O
  Other Names: placebo

SUMMARY:
A Multi-center, Randomized, Double-blind, Parallel Phase Ⅳ Study to Explore the Efficacy of Statin/Choline Fenofibrate Combination Therapy vs Statin Monotherapy in Patients With Inadequately Controlled TG Despite Receiving Statin Monotherapy

ELIGIBILITY:
Inclusion Criteria:

* both male and female who are over 19-year-old
* 200mg/dl≤TG<500mg/dl
* Desired value of LDL-c

  1. very high risk < 70
  2. high risk < 100
  3. moderate risk <130
  4. low risk < 160

Exclusion Criteria:

* patient who is going to have an operation during this study
* patient who has allergy or hypersensitivity of fenofibrate
* patient who has abnormal ECG

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-07-25 (Actual); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
rate of change for Triglyceride based on baseline | 8week

CONTACTS AND LOCATIONS:
Locations (1):
- Hallym University Dongtan Sacred Heart Hospital, Hwaseong-si, South Korea

REFERENCES:
- [Derived] Park MS, Youn JC, Kim EJ, Han KH, Lee SH, Kim SH, Kim BJ, Kwon SU, Ryu KH. Efficacy and Safety of Fenofibrate-Statin Combination Therapy in Patients With Inadequately Controlled Triglyceride Levels Despite Previous Statin Monotherapy: A Multicenter, Randomized, Double-blind, Phase IV Study. Clin Ther. 2021 Oct;43(10):1735-1747. doi: 10.1016/j.clinthera.2021.08.005. Epub 2021 Sep 10. PMID 34518033